CLINICAL TRIAL: NCT04456569
Title: Geniculate Artery Embolization for Osteoarthritis: Pilot Study
Brief Title: Geniculate Artery Embolization for Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAD-2019-27368
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Osteo Arthritis Knee; Arthritis; Osteoarthritis; Osteoarthritis, Knee
Keywords: Embolotherapy
MeSH Terms: conditions — Arthritis; Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- GAE + Standard of Care (Experimental): Participants in this arm will receive geniculate artery embolization and standard of care.
  Interventions: Device: Geniculate Artery Embolization
- Standard of Care (No Intervention): Participants in this arm will receive standard of care only.

INTERVENTIONS:
Device: Geniculate Artery Embolization — All patients within the embolization group will undergo unilateral angiography and embolization of the appropriate treatment limb geniculate arteries. For patients with bilateral disease the more clinically symptomatic side will be chosen as the treatment/control knee.
  Arms: GAE + Standard of Care

SUMMARY:
The need for exploration of more definitive and cost effective non-arthroplasty treatments of osteoarthritis (OA) has been demonstrated by the orthopedic and health economic research.

Embolotherapy of neovessels associated with OA joints has been shown to be promising in patients with knee OA. There is a need for level one evidence drawn from randomized clinical trials to prove the safety, feasibility and efficacy of knee embolotherapy compared to standard of care.

This randomized pilot study will assign 10 patients with mild-moderate OA to undergo geniculate artery embolization plus standard of care (defined in this study as: physical therapy and oral anti-inflammatory medications, with a maximum of 1 joint injection at the time of enrollment) and 10 patients to receive only medical standard of care (also having had a maximum of 1 joint injection prior to enrollment). The goal of this pilot study is to obtain preliminary estimates of safety and efficacy of embolotherapy to provide sustained symptom control and modify disease progression in patients with mild to moderate knee OA.

DETAILED DESCRIPTION:
This is a single center, two-arm, open label, pilot study to assess feasibility and safety and obtain a preliminary estimate of efficacy of geniculate artery embolization in reducing pain compared to a control group undergoing conservative presurgical management. The 20 patients will be randomly divided into two groups of 10 in 1:1 allocation. One group will have embolization of the geniculate artery branches and standard of care while the other will have only the standard care. Following the completion of the 10 participants in each arm, a safety and data review will be undertaken (Visit 4 in the GAE group and Visit 2 of the SOC). The data will be assessed regarding the trends between the groups as they relate to KOOS/WOMAC pain scale, MRI / Xray evaluation of OA, and presence of inflammatory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Between 40 - 70 years of age.
* Unilaterally dominant symptomatic OA (bilateral radiographic OA will not exclude).
* Symptomatically refractory of at least 3 months of medical and/or rehabilitation measures (anti-inflammatory drugs, and/or physical therapy, and/or strength conditioning, and/or intra-articular injections of the affected knee in the last 3 months).
* Kellgren-Lawrence grade 1, 2, or 3 on radiograph of the knee
* Willing to comply with the protocol requirements and willing to undergo non- contrast MRI during screening and at 12 months.
* Willing to comply with regular follow up during the 12 month follow-up period.
* Not a current candidate for partial or total knee arthroplasty.
* WOMAC Score >=6 in at least 2 categories.

Exclusion Criteria:

* BMI >35 kg/m2
* Advanced peripheral arterial disease (resting ABI <= 0.9).
* Known significant peripheral arterial disease precluding common femoral catheterization
* Have smoked tobacco regularly (smoking 1 or more tobacco product(s) per week) within the last year
* Diabetics with hemoglobin A1C of >9%
* Previous lower extremity embolization
* Uncontrolled emotional disorders per patient medical history
* Chronic pain syndrome or currently under a pain contract.
* Anatomic variants involving the lower extremities which would increase the risk of non-target embolization
* Renal insufficiency based on an estimated GFR<45 ml/min who are not already on hemodialysis.
* Abnormal INR (>1.5)
* Platelet count <50x109/L.
* Currently receiving medications for anticoagulation which cannot safely be held for the procedure and for 7 days post-procedure.
* Known severe allergy to iodine which cannot be adequately pre-medicated
* Pregnant or intend to become pregnant within 6 months of the procedure
* Contraindication to drugs used for moderate sedation during interventional procedures, including Midazolam and Fentanyl
* Life expectancy <60 months
* Currently enrolled or who plan to enroll in other investigations that conflict with follow-up testing or confounds data in this trial
* Contraindications to medical and physical rehabilitative treatments of OA.
* Advanced atherosclerosis.
* Current or previous lower extremity fistula.
* Rheumatoid arthritis or seronegative arthropathies.
* WOMAC Pain Scale < 6
* Steroid injection in the affected joint within 3 months of screening. I- n investigator assessment, patient is not a candidate for study participation

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety as Assessed by Grade 3-4 Adverse events | 12 months
  Safety will be reported using the combined number of grade 3 and 4 adverse events that occur in each arm.

SECONDARY OUTCOMES:
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) | baseline, 1 month, 6 months, 12 months
  The KOOS measures 5 patient-relevant dimensions, each scored separately:
  Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items).
  Items are rated on a 5-point Likert scale from 0 (No problems) to 4 (Extreme problems). Dimension scores are calculated as the mean score of the included items divided by 4 and multiplied by 100. Range of subscale scores is 0-100 with higher scores indicating better function.
Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | baseline, 1 month, 6 months, 12 months
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a self-administered questionnaire consisting of 24 items divided into 3 subscales: Pain (5 items), stiffness (2 items), and physical function (17 items). Items are rated on a Likert scale of 0 (extreme) to 4 (none). Raw sub-scale scores are normalized to produce percentage scores in accordance with the KOOS by multiplying each score by 100/96. Total scores are a sum of the normalized sub-scales scores and range 0-100, with higher scores indicating better functioning.
IL-6 Concentration | baseline, 1 month, 12 months
  Interleukin-6 concentrations will be measured in the serum and joint aspirate and reported in units of pg/ml.
Prostaglandin E2 Concentration | baseline, 1 month, 12 months
  Prostaglandin E2 concentrations will be measured in the serum and joint aspirate and reported in units of pg/ml.
Matrix Metalloprotinase 1 Concentration | baseline, 1 month, 12 months
  Matrix Metalloprotinase 1 concentrations will be measured in the serum and joint aspirate and reported in units of ng/ml.
Vascular Endothelial Growth Factor Concentration | baseline, 1 month, 12 months
  Vascular Endothelial Growth Factor concentrations will be measured in the serum and joint aspirate and reported in units of pg/ml.
C-Reactive Protein Concentration | baseline, 1 month, 12 months
  C-Reactive Protein concentrations will be measured in the serum and reported in units of mg/L.
Erythrocyte Sedimentation Rate | baseline, 1 month, 12 months
  Erythrocyte sedimentation rate will be performed using serum and reported in units of mm/hr.

OTHER OUTCOMES:
Feasibility as Assessed by Protocol Adherence | 12 months
  Feasibility will be assessed and reported as the number of participants in each arm who drop out due to a lack of protocol adherence.
Feasibility as Assessed by Recruitment Rate | 12 months
  Feasibility will be assessed and reported as the mean number of participants who are enrolled each month over the length of the study (12 months).

CONTACTS AND LOCATIONS:
Overall Officials: Reza Talaie, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States